CLINICAL TRIAL: NCT04480671
Title: Impact of Level III Support Procedure on Normalization of Enlarged Genital Hiatus After Minimally Invasive Sacrocolpopexy: a Randomized Controlled Trial
Brief Title: Impact of Level III Support Procedure on Enlarged Genital Hiatus After Minimally Invasive Sacrocolpopexy
Acronym: MERIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Stephanie Glass Clark, Assistant Professor of Urogynecology and Reconstructive Pelvic Surgery, Department of Obstetrics, Gynecology and Reproductive Sciences, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19110286
Record Dates: First submitted 2019-12-17; First posted 2020-07-21 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Postoperative pelvic exams measuring anatomic recurrence of pelvic organ prolapse will be performed by a qualified examiner masked to the original surgery randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacrocolpopexy (Other): This group will only receive the sacrocolpopexy for their pelvic organ prolapse repair.
  Interventions: Procedure: Minimally Invasive Sacrocolpopexy; Other: Transperineal ultrasound of the Pelvic Floor
- Sacrocolpopexy and concomitant level III support procedure (Active Comparator): This randomized group will receive an additional vaginal repair for level III support at the conclusion of the sacrocolpopexy.
  Interventions: Procedure: Level III support procedure; Procedure: Minimally Invasive Sacrocolpopexy; Other: Transperineal ultrasound of the Pelvic Floor

INTERVENTIONS:
Procedure: Level III support procedure — A level III support procedure is aimed at repairing the distal support of the vagina with either a posterior colporrhaphy and/or a perineorrhaphy.
  Arms: Sacrocolpopexy and concomitant level III support procedure
Procedure: Minimally Invasive Sacrocolpopexy — All study participants are planning with their surgeon a minimally invasive sacrocolpopexy (robotic or laparoscopic) to repair pelvic organ prolapse.
Other: Transperineal ultrasound of the Pelvic Floor — Subjects from either arm will be invited to participate in this exploratory arm of the study. If they choose to participate, they will have a preoperative ultrasound performed and an ultrasound performed at the time of their 6 month visit.

SUMMARY:
This is a randomized controlled surgical trial evaluating the use of a concomitant posterior colporrhaphy and/or perineorrhaphy at the conclusion of minimally invasive sacrocolpopexy to narrow enlarged genital hiatuses in a population of women with pelvic organ prolapse. The study's primary outcome is the proportion of women at 6 months postoperatively who still have an enlarged genital hiatus.

An exploratory sub-aim (as of October 2021) of the study is to evaluate the levator hiatal area as compared with the genital hiatus by using preoperative and postoperative transperineal ultrasounds. Subjects will be invited to participate, but is not required for study participation.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with pelvic organ prolapse (POP)
* Planning a surgical repair of POP with minimally invasive sacrocolpopexy
* Preoperative resting genital hiatus measure between 4.0 and 7.5cm

Exclusion Criteria: subjects who are unable to complete questionnaires or repeat office exams or if they do not otherwise meet inclusion criteria above

*Note: we will NOT exclude patients based on prior surgical history (including prior posterior colporrhaphy)*

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Enlarged Genital Hiatus at 6 months postoperatively | 6 months postoperatively
  Proportion of subjects with enlarged genital hiatus on pelvic exam

SECONDARY OUTCOMES:
Composite prolapse recurrence | 12 months
  Any anatomic prolapse recurrence beyond the hymen, symptomatic on questionnaire, or retreatment for prolapse with surgery or pessary.
Subjective prolapse recurrence | 24 months
  Any symptomatic recurrence of prolapse on questionnaire
Dyspareunia postoperatively | 6, 12 months postoperatively
  Incidence of pain with sex (dyspareunia), ascertained with the use of a validated questionnaire for sexual function [the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR)].This questionnaire indicates worse pain with sex with higher score.
Sexual Function postoperatively | 6, 12 months postoperatively
  Assessment of sexual function, ascertained with the use of a validated questionnaire for sexual function [the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR)]. This questionnaire helps us determine what impact pelvic organ prolapse has on sexual activity.
Pelvic Floor Distress Inventory Change | baseline, 6, 12 months postoperatively
  Measurement of pelvic floor distress change, using the Pelvic Floor Distress Inventory questionnaire (PFDI-20) which is a validated questionnaire used for pelvic floor disorders and their impact on patient quality of life.
Levator Hiatal Area | baseline, 6 months postoperatively
  Measurement of the levator hiatus on transperineal ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Bradley MS, Askew AL, Vaughan MH, Kawasaki A, Visco AG. Robotic-assisted sacrocolpopexy: early postoperative outcomes after surgical reduction of enlarged genital hiatus. Am J Obstet Gynecol. 2018 May;218(5):514.e1-514.e8. doi: 10.1016/j.ajog.2018.01.046. Epub 2018 Feb 6. PMID 29425837
- [Background] Nosti PA, Umoh Andy U, Kane S, White DE, Harvie HS, Lowenstein L, Gutman RE. Outcomes of abdominal and minimally invasive sacrocolpopexy: a retrospective cohort study. Female Pelvic Med Reconstr Surg. 2014 Jan-Feb;20(1):33-7. doi: 10.1097/SPV.0000000000000036. PMID 24368486
- [Background] Siddiqui NY, Geller EJ, Visco AG. Symptomatic and anatomic 1-year outcomes after robotic and abdominal sacrocolpopexy. Am J Obstet Gynecol. 2012 May;206(5):435.e1-5. doi: 10.1016/j.ajog.2012.01.035. Epub 2012 Feb 1. PMID 22397900
- [Background] Vaughan MH, Siddiqui NY, Newcomb LK, Weidner AC, Kawasaki A, Visco AG, Bradley MS. Surgical Alteration of Genital Hiatus Size and Anatomic Failure After Vaginal Vault Suspension. Obstet Gynecol. 2018 Jun;131(6):1137-1144. doi: 10.1097/AOG.0000000000002593. PMID 29742664
- [Background] Carter-Brooks CM, Lowder JL, Du AL, Lavelle ES, Giugale LE, Shepherd JP. Restoring Genital Hiatus to Normative Values After Apical Suspension Alone Versus With Level 3 Support Procedures. Female Pelvic Med Reconstr Surg. 2019 May/Jun;25(3):226-230. doi: 10.1097/SPV.0000000000000528. PMID 29210807
- [Background] Sutkin G, Zyczynski HM, Sridhar A, Jelovsek JE, Rardin CR, Mazloomdoost D, Rahn DD, Nguyen JN, Andy UU, Meyer I, Gantz MG; NICHD Pelvic Floor Disorders Network. Association between adjuvant posterior repair and success of native tissue apical suspension. Am J Obstet Gynecol. 2020 Feb;222(2):161.e1-161.e8. doi: 10.1016/j.ajog.2019.08.024. Epub 2019 Aug 23. PMID 31449806